CLINICAL TRIAL: NCT06770803
Title: High Versus Low Pneumoperitoneum PressUre for Parenchymal Transection in Minimally Invasive Major Liver Surgery - a Non-inferiority, Multicenter, Randomized, Controlled Trial
Brief Title: High Versus Low Pneumoperitoneum PressUre for Parenchymal Transection in Minimally Invasive Major Liver Surgery
Acronym: PPULS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Collaborators: University of Ulm (Other); University Hospital Dresden (Other); Groeninge Hospital, Kortrijk, Belgium (Unknown)
Responsible Party: Principal Investigator, Arianeb Mehrabi, MD, Professor, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: S-729/2024
Record Dates: First submitted 2024-12-30; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Liver Surgery; Minimal Invasive Surgery; Major Liver Resection
Keywords: Pneumoperitoneum; minimal-invasive liver surgery; intraoperative blood loss
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Intervention Model Description: This trial is a multicenter, randomized, controlled, non-inferiority trial with a two-arm parallel-group design. Patients will be randomized to either the LPP or HPP group during the parenchymal transection phase of MILR. Study interventions include intraoperative measures such as blood sampling, peritoneal biopsies, and liver tissue collection to assess intraoperative tissue damage. Transesophageal echocardiography will be employed to detect CO2 embolisms, while the quality of the surgical field will be evaluated using the Leiden Surgical Rating Scale (L-SRS). Follow-up and data collection involves gathering postoperative data on morbidity, complications, and recovery quality, alongside analyzing blood and biopsy samples for cytokine and molecular markers. The study will also monitor long-term outcomes, including hospital readmission, survival rates, and histopathological findings in cases of malignancy.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Pressure Pneumoperitoneum (Active Comparator): Intraperitoneal insufflation pressures (IIP) during the parenchymal transection phase of liver resection will be different between the two study groups. Baseline IIP of the surgical procedure will be ≤10 mmHg. IIP will be elevated to ≥14 mmHg in the intervention group during the parenchymal transection phase of liver resection.
  Interventions: Procedure: High Pressure Pneumoperitoneum
- Low Pressure Pneumoperitoneum (Sham Comparator): Intraperitoneal insufflation pressures (IIP) during the parenchymal transection phase of liver resection will be different between the two study groups. Baseline IIP of the surgical procedure will be ≤10 mmHg. IIP will be maintained at ≤10 mmHg in the control group.
  Interventions: Procedure: Low Pressure Pneumoperitoneum

INTERVENTIONS:
Procedure: High Pressure Pneumoperitoneum — The objective of this trial is to determine whether the maintenance of a low intraperitoneal insufflation pressure (IIP) of ≤10 mmHg during the parenchymal transection phase of conventional and robotic-assisted laparoscopic liver resection is non-inferior to a higher IIP of ≥14 mmHg in terms of intraoperative blood loss, gas embolisms, perioperative morbidity, and mortality.
  Arms: High Pressure Pneumoperitoneum
Procedure: Low Pressure Pneumoperitoneum — The objective of this trial is to determine whether the maintenance of a low intraperitoneal insufflation pressure (IIP) of ≤10 mmHg during the parenchymal transection phase of conventional and robotic-assisted laparoscopic liver resection is non-inferior to a higher IIP of ≥14 mmHg in terms of intraoperative blood loss, gas embolisms, perioperative morbidity, and mortality.
  Arms: Low Pressure Pneumoperitoneum

SUMMARY:
Minimally invasive techniques in liver surgery gain popularity as they facilitate postoperative recovery while achieving comparable oncologic outcomes to the open approach. No consensus on the application of pneumoperitoneum pressure in minimal invasive liver resections (MILR) has been reached yet, as prospective clinical studies are scarce. The positive pressure of the CO2 pneumoperitoneum reduces intraoperative blood loss during MILR alongside the development of new transection devices and advancements in inflow control. Low-pressure pneumoperitoneum on the other hand has been shown to decrease postoperative pain scores and analgesic consumption in comparison to standard pneumoperitoneum, and international guidelines recommend the application of "the lowest intra-abdominal pressure allowing adequate exposure of the operative field rather than a routine pressure". Nevertheless, evidence for the application of low-pressure pneumoperitoneum is only moderate to low, requiring additional studies to better define its safety. To address this oxymoron, the investigators conduct a randomized non-inferiority trial to investigate the effect of low in comparison to high-pressure pneumoperitoneum during the transection phase of major MILR on intraoperative blood loss while also evaluating the risk of embolic complications.

ELIGIBILITY:
Inclusion Criteria:

* age equal or older than 18 years and
* capacity of consent and
* planned elective conventional laparoscopic or da Vinci-assisted major liver resection or resections near the liver hilum or the hepatic venous vasculature. Major liver resections are defined as the resection of 3 liver segments or more (right and left partial hepatectomies, extended right and left hepatectomies, liver resections of 3 or more segments). Right posterior sectionectomies and mesohepatectomies of ≥2 liver segments are considered resections in proximity to the liver hilum or hepatic venous vasculature.

Exclusion Criteria:

* the participation in another trial with interference of intervention and outcome of this study,
* being a woman who is pregnant or breast-feeding or planning to become pregnant,
* American Society of Anesthesiologists (AS) score >3,
* language barrier,
* any contraindication to a minimal invasive surgical approach or intolerance to pneumoperitoneum
* a patent foramen ovale (PFO) or any other structural cardiac defect that facilitates paradoxical gas embolisms,
* diagnosis of neuromuscular disease, heart failure NYHA > class II or chronic obstructive pulmonary disease (COPD)
* being on oral anticoagulation therapy other than Aspirin 100mg daily or any other condition known to increase the risk of bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Intraoperative blood loss | From the time of randomization until the completion of the liver surgery, assessed up to 24 hours.

SECONDARY OUTCOMES:
Incidence of CO2 embolisms | intraoperative
  Incidence of CO2 embolisms in the right atrioventricular system detected by intraoperative transesophageal echocardiography
Morbidity rate | 90 days postoperative
  Postoperative complication rate
Mortality rate | 90 days postoperative
  Postoperative mortality

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request, the data generated by the current research that supports our future article, would be made available as soon as possible, wherever legally and ethically possible.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Giehl-Brown E, Khajeh E, Dehne S, Czigany Z, Gutzeit O, Neuhaus C, Riediger C, Birgin E, Rahbari N, D'Hondt M, Lurje G, Weigand M, Michalski C, Mehrabi A, Kahlert C. High versus low pneumoperitoneum PressUre for parenchymal transection in minimally invasive major liver surgery (PPULS)-a non-inferiority, multicenter, randomized, controlled trial. Trials. 2025 Dec 1;26(1):556. doi: 10.1186/s13063-025-09269-9. PMID 41327288